CLINICAL TRIAL: NCT00668304
Title: Prospective, Multicenter, Open, Uncontrolled Trial to Evaluate the Time to Bacterial Eradication and Key Symptom Relief in the Treatment of Acute Bacterial Maxillary Sinusitis With Moxifloxacin 400 mg QD
Brief Title: Trial to Evaluate Time to Symptom Relief and Elimination of Infecting Bacteria in Treating Sinusitis With Avelox
Acronym: SPEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100569
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Maxillary Sinusitis
Keywords: Sinusitis
MeSH Terms: conditions — Maxillary Sinusitis; Sinusitis | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Moxifloxacin 400 mg once orally daily

SUMMARY:
This study evaluated the time to bacteriological eradication of common pathogens during moxifloxacin therapy for acute bacterial maxillary sinusitis. The study also examined the time to resolution of key symptoms associated with sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute sinusitis with signs and symptoms present for >7 days but < 28 days as defined by A), radiographic, and B) clinical criteria, as follows:a. The presence of 1 or more of the following on a radiographic paranasal sinus film (Waters' view) or limited CT scan:** evidence of air-fluid levels** opacification. The presence of at least one major and one minor symptom as defined in the list below:** Major Symptoms*** Purulent anterior or posterior nasal discharge*** Unilateral moderate or severe facial pain or malar tenderness** Minor Symptoms*** Cough or frequent throat clearing*** Frontal headache*** Halitosis*** Fever (oral > 38.0°C/100.4°F, tympanic > 38.5°C/101.2°F)*** Purulent secretions obtained via middle meatus secretion sampling using nasal endoscopic technique; the specimen sent for Gram stain, culture and susceptibility testing prior to initiation of antimicrobial therapy

Exclusion Criteria:

* History of chronic sinusitis defined as greater than four weeks of continuous symptoms (patients with history of sinus surgery may be included; patients with recurrent sinusitis may be included)
* Known bacteremia, meningitis or infection infiltrating the tissues neighboring the sinuses- Received systemic antibacterial therapy likely to be effective in sinusitis for more than 24 hours within 7 days of enrollment- A requirement for concomitant systemic antibacterial therapy with agents other than those specified in this protocol- Known immunodeficiency diseases including AIDS (CD4 <200)- On topical nasal or systemic corticosteroids, unless they have been on a stable dose for > 4 weeks prior to enrollment- History of allergy to quinolone antibiotics or related compounds- Pregnant or breast feeding- Of childbearing potential in whom pregnancy cannot be excluded by a negative pregnancy test and who are not using reliable barrier method of contraception
* Received an investigational drug in the past 30 days- Unable to take oral medication- Known to have congenital or sporadic syndromes of QTc prolongation or receiving concomitant medication reported to increase the QTc interval (e.g. amiodarone, sotalol, disopyramide, quinidine, procainamide, terfenadine)
* End stage liver cirrhosis (class Child-Pugh C)- Severe renal impairment requiring dialysis
* Previous history of tendinopathy associated with quinolones- Any symptoms that suggest that the patient's current illness is allergic rhinitis (e.g., repetitive sneezing, itchy nose or eyes, provocation by an allergen) and not acute bacterial sinusitis
* Diagnosis of rapidly fatal illness with a life expectance of less than 6 months- Previously enrolled in this clinical study- Uncorrected hypokalaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2004-06; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Time to bacteriological eradication in those who are microbiologically valid for S. pneumoniae, M. catarrhalis, and H. influenzae | Days 1, 2, 3 of treatment

SECONDARY OUTCOMES:
Patient-reported symptom improvement using SNOT-16 questionnaire | Up to End of Treatment (Day 10-13)
Clinical Response | End of Treatment
Bacteriological Response | End of Treatment
Activity Impairment Assessment questionnaire | Up to End of Treatment (Day 10-13)
Incidence of Premature Termination | Premature Termination
Adverse Events Collection | Up to End of Treatment (Day 10-13)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (34):
- United States (29):
  - Birmingham, Alabama
  - Hoover, Alabama
  - Jonesboro, Arkansas
  - Searcy, Arkansas
  - Fresno, California
  - Riverside, California
  - San Francisco, California
  - Colorado Springs, Colorado
  - Longmont, Colorado
  - Bridgeport, Connecticut
  - DeLand, Florida
  - Shreveport, Louisiana
  - Detroit, Michigan
  - North Massapequa, New York
  - Rochester, New York
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Yukon, Oklahoma
  - Lake Oswego, Oregon
  - Harrisburg, Pennsylvania
  - Greenville, South Carolina
  - Orangeburg, South Carolina
  - Jackson, Tennessee
  - Carrollton, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Winchester, Virginia
  - Spokane, Washington
- Argentina (5):
  - San Juan Bautista, Buenos Aires
  - Buenos Aires, Buenos Aires F.D.
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province